

# Intraoperative case series study: trial rasp position versus SL-PLUS™ MIA Ti/HA femoral hip stem position

Short Title: SL-PLUS™ MIA Ti/HA femoral hip stem 15-4567-03

Statistical Analysis Plan -Final Version-Version: 1.0 (2017/09/21)

## Nondisclosure Statement

This document contains information confidential and proprietary to Smith & Nephew, and is conditionally loaned only. By retention, the recipient agrees not to reproduce or copy it in whole or in part, disclose any or all of its contents without prior written permission, or make any use of it contrary to Smith & Nephew. Recipient further agrees to return it upon request.



# **Contents**

| 1. | Signature page | 4 |
|---|---|---|
| 2. | Revision History | 5 |
| 3. | Acronyms | 5 |
| 4. | Introduction | 5 |
| 5. | Study Objectives | 6 |
| 6. | Investigation Plan | 6 |
| 6.1 | . Study Design | 6 |
| 6.2 | | |
| 6.3 | . Sample Size Determination | 7 |
| 6.4 | . Visit Schedule and Visit Window | 8 |
| 6.5 | . Primary Endpoint Evaluation | 8 |
| 6.6 | . Secondary Endpoints Evaluations | 9 |
| 6.7 | . Safety | 9 |
| 7. | Statistical Methods | 9 |
| 7.1 | . General Reporting Conventions | 9 |
| 7.2 | . Study Populations | 10 |
| 7.3 | . Adjustments for Interim Analyses and Multiple Endpoints | 10 |
| 8. | Statistical Methods and Evaluations | 10 |
| 8.1 | . Subject Disposition and Accountability | 10 |
| 8.2 | . Demographic and Baseline Characteristics | 11 |
| 8.3 | . Treatment Administration | 11 |
| 8.4 | . Effectiveness Evaluations | 11 |
| 8 | 3.4.1. Primary Analysis | 11 |
| 8.5 | . Safety Evaluations | 12 |
| 8 | 3.5.1. Adverse Events, Serious Adverse Events and Device Deficiency | 12 |
| 8 | 3.5.2. Radiographic Data | 12 |
| 8.6 | . Other Evaluations | 12 |
| 9. | Changes to Planned Analyses | 12 |
| 10. | References | 12 |
| 11. | List of Tables | 12 |
| 12. | Appendix | 15 |



| 12.1. | Inclusion/Exclusion & Informed Consent | 15 |
|-------|----------------------------------------|----|
| 12.2. | Demographics | 15 |
| 12.3. | Pre-Operative Analysis | 18 |
| | Operative Analysis | |
| 12.5. | Independent Image Review Fluoroscopy | 26 |
| 12.6. | Device Deficiency | 27 |
| 12.7. | Adverse Event Form | 28 |
| 12.8. | Serious Adverse Event Report Form | 30 |
| 12 9 | End of Study | 32 |



# 1. SIGNATURE PAGE

| Study Title: | Intraoperative case series study: trial rasp position versus SL-PLUS™ MIA Ti/HA femoral hip stem position |
|---|---|
| Study Number: | 15-4567-03 |
| Product: | SL-PLUS™ MIA Ti/HA |
| Report Date: | 21-Sep-2017 |

| Position | Signature | Date Approved |
|-----------------------------------------------|-----------|---------------|
| Fiona Schlomowitsch<br>Clinical Study Manager | +Mon f | 28-Sep-2017 |
| Nick Bornschein<br>Biostatistician STATWORX | | 16-Oct-2017 |
| Alan Rossington Reviewing Biostatistician | Alloringh | 12-Oct-2017 |



# 2. REVISION HISTORY

| Version<br>Number | Reason for Change or Change Control<br>Number | Document Author |
|---|---|---|
| 0.1 | Initial Draft Version | Nick Bornschein |
| 0.2 | Draft Version | Nick Bornschein |
| 0.3 | Draft Version | Nick Bornschein |
| 0.4 | Draft Version | Nick Bornschein |
| 0.5 | Draft Version | Nick Bornschein |
| 0.6 | Draft Version | Nick Bornschein |
| 0.7 | Draft Version | Nick Bornschein |
| 0.8 | Draft Version | Nick Bornschein |
| 0.9 | Draft Version | Nick Bornschein |
| 1.0 | Final Version | Nick Bornschein |

## 3. ACRONYMS

Table 1: Acronyms

| Acronyms | Term |
|-----------------|--------------------------------|
| ADE | Adverse Device Effects |
| AE | Adverse Event |
| CI | Confidence Interval |
| CRF | Case Report Form |
| DD | Device Deficiency |
| FAS | Full Analysis Set |
| m <sub>50</sub> | Median |
| Max | Maximum |
| Min | Minimum |
| MRT | Multiple Response Table |
| N | Available Records (count) |
| SADE | Serious Adverse Device Effects |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| THA | Total Hip Arthroplasty |

## 4. INTRODUCTION

With an increasing life expectancy, the demand of total hip arthroplasties is rising while the success of the hip implant depends to the position of the femoral stem. The correct position of a cemented hip stem is planned preoperatively. During surgery, the final



position of the rasp should correspond to the preoperatively determined position and the same position should be adopted by the cemented femoral stem.

The SL-PLUS™ MIA Ti/HA femoral hip stem study is going to evaluate the difference between the final position of the stem and the last trial rasp.

#### 5. STUDY OBJECTIVES

The study objective is to evaluate if there is a difference between the femoral position of the last trial rasp and the final implant position of the SL-PLUS™ MIA Ti/HA femoral hip stem.

## **Primary Endpoint:**

The primary endpoint is the mean difference D between the position of the last trial rasp and the final implant position of the SL-PLUS™ MIA Ti/HA femoral hip stem. The difference D is determined by analyzing standardized fluoroscopic images taken during surgery.

The difference D is given in mm and is defined as D = x1 - x2 with x1 being the distance between the shoulder of the trial rasp and the tip of the greater trochanter and x2 being the distance between the shoulder of the implant and the tip of the greater trochanter.

The study hypothesis is defined as:

 $H_0$ : The null hypothesis is that there is no mean difference between the position of the last trial rasp and the final implant position of the SL-PLUS<sup>TM</sup> MIA Ti/AH femoral hip stem.

 $H_1$ : The alternative hypothesis is that there is a mean difference between the position of the last trial rasp and the final implant position of the SL-PLUS<sup>TM</sup> MIA Ti/AH femoral hip stem.

# **Secondary Endpoints:**

The secondary endpoints include a measurement of leg length discrepancy preoperatively and after insertion of the SL-PLUS™ MIA Ti/HA femoral hip stem. In addition, intraoperative complications will be collected.

#### 6. INVESTIGATION PLAN

## **6.1. STUDY DESIGN**

This is an observational, single arm, prospective, multi-center, case series study to collect intraoperative data from 40 subjects implanted with the SL-PLUS™ MIA Ti/HA femoral hip stem at 4 sites in Europe.

Data from eligible subjects, who have provided written and informed consent for the collection of their coded data, will be recorded on specially designed case report forms (CRFs).



No follow-up visits after surgery is planned for study participants. Therefore, total study duration for study participants is completed with surgery.

A final data analysis describing the study outcome is planned after completion of study assessments.

#### 6.2. RANDOMIZATION PLAN

No randomization algorithm was followed for patient recruitment.

#### **6.3. SAMPLE SIZE DETERMINATION**

The following hypotheses will be tested:

 $H_0$ : The null hypothesis is that there is no mean difference between the position of the last trial rasp and the final implant position of the SL-PLUS<sup>TM</sup> MIA Ti/AH femoral hip stem.

 $H_1$ : The alternative hypothesis is that there is a mean difference between the position of the last trial rasp and the final implant position of the SL-PLUS<sup>TM</sup> MIA Ti/AH femoral hip stem.

$$H_0$$
:  $\mu = 0 \ vs. H_1$ :  $\mu \neq 0$ 

In 2007, a non-published cadaver test was performed to measure the difference D between the position of the last trial rasp and the implant position of the SL-PLUS<sup>TM</sup> MIA Ti/AH femoral hip stem. A total of 4 femoral hip stems were implanted into the cadaveric femur. The range of the measured difference was found to be between 0mm and 6mm. However, it is most likely that the maximum difference will be greater 6mm when more cases are studied. To compensate for the small number of evaluated cases, the anticipated variation in D will be extended to 10mm with an estimated standard deviation of 2.5mm. A correlation  $\rho$  between the distances  $\kappa_1$  and  $\kappa_2$  is certainly positive but it is unknown how strong the correlation is. The standard deviation sd of the difference D has the following relationship with the standard deviations  $\kappa_1$  and  $\kappa_2$  for distances  $\kappa_1$  and  $\kappa_2$ :

$$sd^2 = sd_1^2 + sd_2^2 - 2 \rho sd_1 sd_2$$

Since  $\rho>0$  and assuming that  $\rho=0$  will lead to a larger sd and therefore a larger sample size. If assumed that  $sd_1=sd_2$ , then  $sd^2=2sd_1^2$ . So assuming  $sd_1$  and  $sd_2$  being equal, the sd will also lead to a larger sample size. Therefore, assuming that the correlation is zero and allowing for both standard deviations  $sd_1$  and  $sd_2$  to be 2.5mm is a conservative approach for computing sample size.

According to orthopaedic surgeons, the maximum difference between the position of the rasp and implant without clinical significance is considered to be 2mm. The standard deviations of  $sd_1$  and  $sd_2$  are estimated as approximately 2.5mm estimated based on the assumptions above and data for the range of difference.

The sample size calculation is based on a two-sided test. The significance level and power of the study are chosen to be 0.05 and 0.90; the minimum mean difference  $\Delta$  is identified as 2 mm; the standard deviations  $sd_1$  and  $sd_2$  are 2.5mm; the correlation between  $x_1$  and  $x_2$  is set to 0. The following formula can be used to calculate the sample size:



$$N \geq \frac{2(T_{N-1,\alpha/2} + T_{N-1,\beta})^2 s d^2}{\Delta^2}$$

The SAS POWER procedure is used to compute the sample size and at least 35 subjects are needed for the study.

# 6.4. VISIT SCHEDULE AND VISIT WINDOW

Table 1 shows the evaluations completed at each visit.

**Table 2: Visit Schedule** 

| Study Visit<br>Schedule | Pre-Operative | Surgery<br>Peri-<br>Operative |
|---|---|---|
| Patient Information and Informed Consent | x | |
| Inclusion/Exclusion<br>Criteria | x | |
| Demographics/Medical<br>History | x | |
| Radiographic assessment | x | |
| Operative Data<br>Collection | | x |
| Fluoroscopic assessment | | x |
| Measurement of leg length discrepancy | x | x |
| Adverse Event<br>Assessment | <b>x</b> * | x |
| End of Study/Exit | | x |

<sup>\*</sup> if applicable

# **6.5. PRIMARY ENDPOINT EVALUATION**



Once a subject has completed the informed consent procedure and signed the Informed Consent Form (ICF)<sup>1</sup>, the Principal Investigator (PI) or delegated study research staff can complete the screening process with the subject. All potential subjects who undergo the screening process will be documented on a Screening and Enrollment Log, on which reasons for exclusion from or denial to participate should be noted. The primary endpoint analysis of the mean difference D between the position of the last trial rasp and the final implant position of the SL-PLUS<sup>TM</sup> MIA Ti/HA femoral hip stem will be based on full analysis set (FAS) population. The FAS population includes all subjects implanted with a SL-PLUS<sup>TM</sup> MIA Ti/HA femoral hip stem device in combination with a Smith & Nephew cup with consecutive enrollments to the study. Subjects being a screen failure (CRF plate 99, question 1. Screen Failue Yes) will be excluded from the FAS.

A primary endpoint analysis of a sub-group might be performed excluding subjects with low image quality as per defined image review criterias (e.g. trochanter not visible). This depends on the assessment of the independent Image Reviewer.

#### 6.6. SECONDARY ENDPOINTS EVALUATIONS

The secondary endpoint analysis of measurement of leg length discrepancy preoperatively and after insertion of the SL-PLUS™ MIA Ti/HA femoral hip stem (and in addition, collecting intraoperative complications) will also be based on full analysis set (FAS) population.

#### **6.7. SAFETY**

Safety evaluations include the listing of Adverse Events (AE), Serious Adverse Events (SAE), Adverse Device Effects (ADE) and Serious Adverse Device Effects (SADE).

Additionally, listings about Device Deficiency (DD) will be reported.

#### 7. STATISTICAL METHODS

#### 7.1. GENERAL REPORTING CONVENTIONS

Analyses will be generated using Stata version 15.0 or higher.

General summary statistics for <u>numeric data</u> include the available records (N), the mean (Mean), the standard deviation (SD), the median  $(m_{50})$ , the minimum (Min), and the maximum (Max) value. Summary statistics can also be grouped by all relevant categorical variables, for example between lateral / standard or Pre-Op / Surgery/Peri-Op.

For <u>categorical data</u>, the count / available records (N) and percent (%) of data will be presented with the percent based on the number of subjects within the data. Additionally, bar charts will be provided.

<sup>&</sup>lt;sup>1</sup> To eliminate the potential for selection bias, Investigators should consecutively pre-screen all subjects undergoing THA with the SL-PLUS™ MIA Ti/HA femoral hip stem. In order to do so, only the existing information obtained per standard routine medical procedures will be used. No study-specific screening procedures, activities or questionnaires will be performed during pre-screening.



For <u>missing data</u>, a complete accountability report, along with the explanation for lost-to-follow-up, death, revision and withdrawn subjects, is to be provided in the study report. No other adjustment or imputations will be made for missing data.

<u>Multiple response</u> answers (marked with "check all that apply") offer several ways to determine the number of valid observations. By default, all cases with at least one valid response are taken into account. All other observations are treated as missing. Furthermore, one might want to consider cases with complete information only and neglect all cases with one or more missing values (Stata option "casewise"). The results will be provided as multiple response table (MRT).

For any <u>two-group comparison</u>, a paired or unpaired t-Test (depending on the data) will be performed. All t-Tests will be fitted using Stata "ttest" command. No 2+ group comparison is planned in this study, so no baseline must be chosen.

If not mentioned otherwise, all results are reported as a two-sided significance test. Significance values of less than 5% (p < 0.05) are considered as statistically significant. Any confidence intervals (CI) will be based on 95% CIs.

#### 7.2. STUDY POPULATIONS

All subjects who meet the study inclusion and exclusion criteria will be included in the statistical analysis. Subjects being a screen failure as documented on "End of Study" – CRF (plate 99) (answer "yes") will be excluded from the statistical analysis. Statistical analyses will be conducted for demographics, pre-operative information, surgical information and safety data. Demographics will include, but not limited to, gender, age, weight and height. Pre-operative information and surgical information will include any data collected as defined in this protocol. Safety data will include adverse events, serious adverse event, adverse device effect, serious adverse device effect, unanticipated serious adverse device effect, and device deficiency.

Descriptive statistics for continuous variables will include mean, median, minimum, maximum, standard deviation, and 95% confidence interval, if appropriate. Descriptive statistics for discrete variables will include count and percentage.

Subgroup analyses will be provided if they are necessary. The following sections define the details of primary endpoint and secondary endpoints analyses.

## 7.3. ADJUSTMENTS FOR INTERIM ANALYSES AND MULTIPLE ENDPOINTS

No interim analyses are planned and no adjustments will be made for multiple endpoints. Testing for secondary measures is provided as an aid in interpreting study results and no specific claims are being sought based on secondary measures.

#### 8. STATISTICAL METHODS AND EVALUATIONS

## **8.1. SUBJECT DISPOSITION AND ACCOUNTABILITY**

Summaries of subject disposition information will be provided and will include the number of subjects screened, enrolled and completed overall and by site (FAS population), the



number of subjects with data by time point and site (theoretical due), deaths, stem revisions, the expected number (expected) and the number of subjects completing the study (actual and %).

Table 3: Subject Disposition by screening and enrollment

| | N |
|-----------|---|
| Screened | |
| Enrolled | |
| Completed | |
| Total | |

#### 8.2. DEMOGRAPHIC AND BASELINE CHARACTERISTICS

Demographic characteristics including age at surgery, gender, operated study hip side and bilateral subjects, will be listed. Height and weight at surgery will be listed for all subjects who allowed use of this information. All pre-operative observations will be summarized descriptively. Summaries for demographic characteristics will be provided in total and by femoral stem type.

Additionally, pre-operative outcome information will be listed as frequency table and all "other" outcomes will be listed separately.

All tables are provided in the appendix, chapter .

## 8.3. TREATMENT ADMINISTRATION

Implant information of SL-PLUS™ MIA Ti/HA will be summarized descriptively including the operated side (left or right) and use of lateral or standard stem. A graph will show the use of lateral and standard stem per site by gender.

#### **8.4. EFFECTIVENESS EVALUATIONS**

#### 8.4.1. Primary Analysis

If the difference between  $x_1$  and  $x_2$  measured from fluoroscopic images approximately follows a normal distribution, then a two-sided paired T test will be used to test the mean. The test statistic is a t-score defined by the following equation:

$$T = \frac{\overline{D}}{\frac{Sd}{\sqrt{N}}}$$
, where  $\overline{D} = N^{-1} \sum_{N=1}^{i=1} (x_{i1} - x_{i2})$ , and  $Sd = \sum_{i=1}^{N} \frac{(x_1 - D^2)^2}{N-1}$  with  $x_i = x_{i1} - x_{i2}$ ;  $i = 1, \dots N$ 

If the difference does not follow a normal distribution, then the signed rank test will be used to test the hypothesis.



#### 8.5. SAFETY EVALUATIONS

## 8.5.1. Adverse Events, Serious Adverse Events and Device Deficiency

Definitions for safety reporting are outlined in chapter 8.1 of the study protocol and in chapter 6.7 of this document.

General and local intra- and post-operative observations will be summarized as frequency tables.

An overall summary of AEs will be provided including the number and percent of subjects with any AE, any related (definitely, probably, possible) AE, any severe AE, any severe and related AE, any AE resulting in death, and any AE resulting in removal or revision of component(s).

All AE will be summarized with count and percent, such as:

- Category of AE (medical diagnosis)
- Severity
- Relationship to study device and procedure
- Outcome
- Study participation
- Actions taken (multiple response)
- Seriousness

If the AE is serious (SAE), a frequency table of SAE categories will be provided.

A device deficiency is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labelling.

## 8.5.2. Radiographic Data

There are no radiographic data.

#### **8.6. OTHER EVALUATIONS**

There are no other evaluations.

## 9. CHANGES TO PLANNED ANALYSES

No changes were made to planned analyses as outlined in the protocol.

## 10. REFERENCES

None.

#### 11. LIST OF TABLES



**Table 4: Table of Tables** 

| | Tables within the Analysis Plan |
|---|---|
| Table 1 | Acronyms |
| Table 2 | Visit Schedule |
| Table 3 | Subject Disposition by screening and enrollment |
| Table 4 | Table of Tables |
| 12 | .1. Inclusion/Exclusion & Informed Consent |
| Table 5 | Enrollment Eligibility |
| | 12.2. Demographics |
| Table 6 | Age, Height and Weight by Subject |
| Table 7 | Age, Height and Weight by Hip |
| Table 8 | Gender |
| Table 9 | Study Side |
| Table 10 | Bilateral Subject Identification |
| 12.3. Pre-Operative Analysis | |
| Table 11 | Preoperative Planning |
| Table 12 | Planned Stem Size |
| Table 13 | Planned and used Stem Size |
| Table 14 | Planned Stem Type |
| Table 15 | Planned and used Stem Type |
| Table 16 | Diagnostic Reason for THA |
| Table 17 | Dorr Classification of Femoral Bone Typ |
| 12.4. Operative Analysis | |
| Table 18 | Fluoroscopic images done |
| Table 19 | Surgical Approach I |
| Table 20 | Surgical Approach II |
| Table 21 | Type of rasping instrument |
| Table 22 | Implanted Components |



| Table 23 | Implanted Components |
|---|---|
| | Implanted Components |
| Table 25 | Correction of final stem position necessary |
| Table 26 | Leg Length Discrepancy |
| Table 27 | Patient Length Difference |
| 12 | 12.5. Independent Image Review Fluoroscopy |
| Table 28 | Trial rasp analysis |
| Table 29 | Implant analysis |
| Table 30 | Analysis of Distances |
| | 12.6. Device Deficiency |
| Table 31 | Device Deficiency related to an AE |
| Table 32 | Timing of Deficiency |
| Table 33 | Duration, if inter-operative delay occurred |
| Table 34 | List of Deficiency |
| 12.7. Adverse Event Form | |
| Table 35 | List of Adverse Events |
| Table 35 Table 36 | List of Adverse Events Duration of resolved events |
| Table 36 | Duration of resolved events |
| Table 36 Table 37 | Duration of resolved events Severity |
| Table 36 Table 37 Table 38 | Duration of resolved events Severity Relationship to study device and procedure |
| Table 36 Table 37 Table 38 Table 39 | Duration of resolved events Severity Relationship to study device and procedure Serious |
| Table 36 Table 37 Table 38 Table 39 Table 40 | Duration of resolved events Severity Relationship to study device and procedure Serious Actions Taken |
| Table 36 Table 37 Table 38 Table 39 Table 40 Table 41 Table 42 | Duration of resolved events Severity Relationship to study device and procedure Serious Actions Taken Outcome |
| Table 36 Table 37 Table 38 Table 39 Table 40 Table 41 Table 42 | Duration of resolved events Severity Relationship to study device and procedure Serious Actions Taken Outcome Study participation discontinued due to event |
| Table 36 Table 37 Table 38 Table 39 Table 40 Table 41 Table 42 | Duration of resolved events Severity Relationship to study device and procedure Serious Actions Taken Outcome Study participation discontinued due to event 12.8. Serious Adverse Event Report Form |
| Table 36 Table 37 Table 38 Table 39 Table 40 Table 41 Table 42 Table 42 | Duration of resolved events Severity Relationship to study device and procedure Serious Actions Taken Outcome Study participation discontinued due to event 12.8. Serious Adverse Event Report Form SAE |



| | 12.9. End of Study |
|----------|---------------------|
| Table 47 | Screen Failure |
| Table 48 | Completion of study |
| Table 49 | Comments |

# 12. APPENDIX

# 12.1. INCLUSION/EXCLUSION & INFORMED CONSENT

**Table 5: Enrollment Eligibility** 

| Eligibility criteria | Total<br>N = xx |
|----------------------|-----------------|
| No | |
| Yes | |
| If no, reason | |

# 12.2. DEMOGRAPHICS

Table 6: Age, Height and Weight by Subject

| Variable | Statistic | Total*<br>N = xx |
|------------|-----------|------------------|
| | N | |
| | Mean | |
| Age at | Min | |
| surgery | Max | |
| (in years) | SD | |
| | -95% CI | |
| | +95% CI | |
| Height | N | |



| (in cm) | Mean |
|-------------------|---------|
| | Min |
| | Max |
| | SD |
| | -95% CI |
| | +95% CI |
| | N |
| | Mean |
| VA/ a i a da 4 | Min |
| Weight<br>(in kg) | Max |
| | SD |
| | -95% CI |
| | +95% CI |
| | N |
| | Mean |
| | Min |
| ВМІ | Max |
| | SD |
| | -95% CI |
| | +95% CI |

Table 7: Age, Height and Weight by Hip

| Variable | Statistic | Total<br>N = xx |
|------------|-----------|-----------------|
| | Ν | |
| Age at | Mean | |
| surgery | Min | |
| (in years) | Max | |
| | SD | |



| | -95% CI |
|-------------------|---------|
| | +95% CI |
| | N |
| | Mean |
| | Min |
| Height (in cm) | Max |
| ( | SD |
| | -95% CI |
| | +95% CI |
| | N |
| | Mean |
| Weight<br>(in kg) | Min |
| | Max |
| (9) | SD |
| | -95% CI |
| | +95% CI |
| | N |
| | Mean |
| | Min |
| ВМІ | Max |
| | SD |
| | -95% CI |
| | +95% CI |

Table 8: Gender

| Gender | Total<br>N = xx (%) |
|--------|---------------------|
| Female | |
| Male | |



Table 9: Study Side

| Study Side | Total<br>N = xx (%) |
|------------|---------------------|
| Left | |
| Right | |

**Table 10: Bilateral Subject Identification** 

| Contralateral hip enrolled | Total<br>N = xx (%) |
|----------------------------|---------------------|
| No | |
| Yes | |
| If yes, Subject ID | |

# 12.3. PRE-OPERATIVE ANALYSIS

**Table 11: Preoperative Planning** 

| | Statistic | Total<br>N = xx |
|------------|-----------|-----------------|
| | Mean | |
| | Min | |
| Distance X | Max | |
| Distance X | SD | |
| | -95% CI | |
| | +95% CI | |

**Table 12: Planned Stem Size** 

| Stem Size | Total<br>N = xx (%) |
|-----------|---------------------|
| 01 | |
| 00 | |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| 7 | |

Table 13: Planned and used Stem Size

| | Planned Stem Size | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Used Stem Size | 01 | 00 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | Total<br>N = xx (row %) |
| 01 | | | | | | | | | | |
| 00 | | | | | | | | | | |
| 1 | | | | | | | | | | |
| 2 | | | | | | | | | | |
| 3 | | | | | | | | | | |
| 4 | | | | | | | | | | |
| 5 | | | | | | | | | | |
| 6 | | | | | | | | | | |
| 7 | | | | | | | | | | |
| Total<br>N = xx (row %) | | | | | | | | | | |



**Table 14: Planned Stem Type** 

| Stem Type | Total<br>N = xx (%) |
|-----------|---------------------|
| Standard | |
| Lateral | |

Table 15: Planned and used Stem Type

| | Planned Stem Type | | |
|---|---|---|---|
| Used Stem<br>Type | Standard | Lateral | Total<br>N = xx<br>(row %) |
| Standard | | | |
| Lateral | | | |
| Total | | | |
| N = xx<br>(row %) | | | |

**Table 16: Diagnostic Reason for THA** 

| Reasons for THA | Total<br>N = xx (%) |
|-----------------------------|---------------------|
| Osteoarthritis | |
| Rheumatoid Arthritis | |
| Post-Traumatic<br>Arthritis | |
| Avascular Necrosis | |
| Dysplasia | |
| Fracture | |
| Other | |
| If other, specify | |



| 7 |
|-----|
| - 1 |
| - 1 |

**Table 17: Dorr Classification of Femoral Bone Typ** 

| Reasons for THA | Total<br>N = xx (%) |
|-----------------|---------------------|
| Type A | |
| Type B | |
| Type C | |

# 12.4. OPERATIVE ANALYSIS

Table 18: Fluoroscopic images done

| Fluoroscopic images | Total<br>N = xx (%) |
|---------------------|---------------------|
| No | |
| Yes | |

Table 19: Surgical Approach I

| Surgical Approach I | Total<br>N = xx (%) |
|---------------------|---------------------|
| Anterolateral | |
| Posterolateral | |
| Anterior | |
| Other | |
| If other, specify | |



Table 20: Surgical Approach II

| Surgical<br>Approach II | Total<br>N = xx (%) |
|-------------------------|---------------------|
| Standard | |
| Minimal<br>Invasive | |

**Table 21: Type of rasping instrument** 

| Rasping instrument | Total<br>N = xx (%) |
|-------------------------|---------------------|
| Slap Hammer | |
| Woodpecker | |
| Mallet | |
| Combination | |
| If combination, specify | |

Table 22: Implanted Components: Femoral Head

| Femoral Head Typ | Total<br>N = xx (%) |
|-------------------------------------|---------------------|
| Ceramic Ball heads,<br>Biolox delta | |
| Ceramic Ball heads,<br>Biolox forte | |
| CoCr femoral head | |
| Other | |
| Femoral Head Size | Total<br>N = xx (%) |
| 28 | |
| 32 | |



| 36 |
|----|

Table 23: Implanted Components: Acetabular Cup

| Acetabular Cup<br>Type | Total<br>N = xx (%) |
|------------------------------------|---------------------|
| R3™ NO HOLE<br>Acetabular Shells | |
| R3 NO HOLE HA<br>Acetabular Shells | |
| R3 THREE HOLE<br>Acetabular Shells | |
| R3 MULTI HOLE<br>Acetabular Shells | |
| Other | |
| Acetabular Cup Size | Total<br>N = xx (%) |
| 28 | |
| 46 | |
| 48 | |
| 50 | |
| 52 | |
| 54 | |
| 56 | |
| 58 | |
| 60 | |

**Table 24: Implanted Components: Acetabular Liner** 

| Acetabular Liner | Total |
|-------------------------------|------------|
| Type | N = xx (%) |
| R3™ XLPE<br>Acetabular Liners | |



| R3™ INTL Delta<br>Ceramic Liners | |
|----------------------------------|---------------------|
| Acetabular Liner<br>Size | Total<br>N = xx (%) |
| 28 | |
| 32 | |
| 36 | |

Table 25: Correction of final stem position necessary

| Necessity of correction | Total<br>N = xx (%) |
|---|---|
| No | |
| Yes | |
| If yes, method | |
| Smaller ball head<br>length | |
| Larger ball head<br>length | |
| Removal of stem and<br>enlargement of<br>femoral bed with last<br>trial rasp | |
| Other method | |
| If other, specify | |

**Table 26: Leg Length Discrepancy** 

| Log Longth Discrenancy | PreOP | PostOP <sup>2</sup> |
|------------------------|------------|---------------------|
| Leg Length Discrepancy | N = xx (%) | N = xx (%) |

<sup>&</sup>lt;sup>2</sup> CRF: Operative Analysis



| None | | | |
|---|---|---|---|
| Ipsilateral Lo | onger | | |
| Ipsilateral St | norter | | |
| If Ipsilate<br>Longer/Sho | | PreOP<br>N = xx (%) | PostOP <sup>3</sup><br>N = xx (%) |
| | Mean | | |
| | Min | | |
| Ipsilateral | Max | | |
| Longer (mm) | SD | | |
| | -95% CI | | |
| | +95% CI | | |
| | | PreOP | PostOP <sup>4</sup> |
| | | N = xx (%) | N = xx (%) |
| | Mean | | |
| | Min | | |
| lpsilateral<br>Shorter (mm) | Max | | |
| | SD | | |
| | -95% CI | | |
| | +95% CI | | |

**Table 27: Patient Length Difference** 

| Patient ID | lateral /<br>standard | PreOp<br>Leg Length<br>Difference<br>mm | PostOp Leg<br>Length<br>Difference<br>mm |
|---|---|---|---|

<sup>&</sup>lt;sup>3</sup> CRF: Operative Analysis <sup>4</sup> CRF: Operative Analysis



# 12.5. INDEPENDENT IMAGE REVIEW FLUOROSCOPY

Table 28: Trial rasp analysis

| | Statistic | Trial Rasp<br>Analysis<br>N = xx |
|------------------|-----------|----------------------------------|
| | Mean | |
| | Min | |
| <b>-</b> 1. | Max | |
| Distance X1 (mm) | SD | |
| | -95% CI | |
| | +95% CI | |

Table 29: Implant analysis

| | Statistic | Implant<br>Analysi<br>s<br>N = xx |
|-------------|-----------|-----------------------------------|
| | Mean | |
| | Min | |
| Distance X2 | Max | |
| (mm) | SD | |
| | -95% CI | |
| | +95% CI | |

Table 30: Analysis of Distances

| Distance | Mean | Difference | Significance |
|--------------------|------|------------|--------------|
| X1<br>(Trial Rasp) | | | |
| X2<br>(Implant) | | | |



- Graph with Stem Comparison -

# 12.6. DEVICE DEFICIENCY

Table 31: Device Deficiency related to an AE

| Relation to AE | Total<br>N = xx (%) |
|---|---|
| No | |
| Yes | |
| If no, if intervention<br>not made, could<br>have let to SADE | |
| No | |
| Yes | |

**Table 32: Timing of Deficiency** 

| Timing | Total<br>N = xx (%) |
|-----------------------|---------------------|
| Before use | |
| During procedural use | |
| After use | |

Table 33: Duration, if inter-operative delay occurred

| Variable | Statistic | Total<br>N = xx |
|------------------------------------------------|-----------|-----------------|
| | Mean | |
| | Min | |
| Duration of inter-<br>operative delay<br>(min) | Max | |
| | SD | |
| | -95% CI | |
| | +95% CI | |

**Table 34: List of Deficiency** 



# 12.7. ADVERSE EVENT FORM

**Table 35: List of Adverse Events** 

| Description of AE | Total<br>N = xx (%) |
|-------------------|---------------------|

**Table 36: Duration of resolved events** 

| Description of AE | Start Date | End Date |
|-------------------|------------|----------|

**Table 37: Severity** 

| Severity | Total<br>N = xx (%) |
|----------|---------------------|
| Mild | |
| Moderate | |
| Severe | |



Table 38: Relationship to study device and procedure

| | to study<br>device | to study procedure |
|--------------|--------------------|--------------------|
| Relationship | Total | Total |
| | N = xx (%) | N = xx (%) |
| Unrelated | | |
| Possible | | |
| Definite | | |

**Table 39: Serious** 

| Serious | Total<br>N = xx (%) |
|-----------------|---------------------|
| No | |
| Yes | |
| If yes, specify | |
| Anticipated | |
| Unanticipated | |

**Table 40: Actions Taken** 

| None | Total<br>N = xx (%) |
|------------------------------|---------------------|
| Yes | |
| Rest | |
| Yes | |
| <b>Medication Therapy</b> | |
| Yes | |
| Surgery/Procedure | |
| Yes | |
| Removal or revision surgery | |
| Yes | |
| Hospitalization or prolonged | |

| Yes |
|-------------------|
| Other |
| Yes |
| If other, specify |

Table 41: Outcome

| Outcome | Total<br>N = xx (%) |
|----------------------------|---------------------|
| Recovered/Resolved | |
| Resolved with sequelae | |
| Recovering/Resolving | |
| Not recovered/Not resolved | |
| Fatal | |
| Unknown | |

Table 42: Study participation discontinued due to event

| Participation discontinued | Total<br>N = xx (%) |
|----------------------------|---------------------|
| No | |
| Yes | |

# 12.8. SERIOUS ADVERSE EVENT REPORT FORM

Table 43: SAE

| Description of SAE | Total<br>N = xx (%) |
|--------------------|---------------------|



**Table 44: Hospitalization** 

| Hospitalization | Total<br>N = xx (%) |
|-----------------|---------------------|
| Yes | |
| No | |
| Admission Date | |
| Known | |
| Unknown | |
| Discharge Date | |
| Known | |
| Unknown | |

**Table 45: Discharge Date (Duration of hospitalization)** 

| Discharge Date (Duration in days) | Total<br>N = xx (%) |
|-----------------------------------|---------------------|
| Mean | |
| Min | |
| Max | |
| SD | |
| -95% CI | |
| +95% CI | |

Table 46: Involvement of study region

| Study region | Total<br>N = xx (%) |
|--------------|---------------------|
| No | |
| Yes | |



# 12.9. END OF STUDY

Table 47: Screen Failure

| Screen Failure | Total<br>N = xx (%) |
|----------------|-------------------------|
| No | |
| Yes | Excluded from analysis. |
| If yes, reason | |

**Table 48: Completion of study** 

| Completed | Total<br>N = xx (%) |
|---|---|
| Yes | |
| No | |
| If no, reason | |
| Subject withdrew consent after study treatment | |
| Subject not able to return | |
| Subject lost to follow-<br>up after contact<br>attempts were made<br>according to protocol | |
| Investigator judgement | |
| Sponsor terminated study | |
| Subject deceased | |



# **Table 49: Comments**

| Comment |
|---------|